CLINICAL TRIAL: NCT04128956
Title: Aspirin® Plus Rivaroxaban Versus Rivaroxaban Alone for the Prevention of Venous Stent Thrombosis in Patients With Post-thrombotic Syndrome a Multi-center, International, Randomized, Open Label, Controlled Trial
Brief Title: Aspirin® Plus Rivaroxaban Versus Rivaroxaban Alone for the Prevention of Venous Stent Thrombosis in Patients With PTS
Acronym: ARIVA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recommendation by DSMB
Sponsor: University of Zurich (Other)
Collaborators: University Hospital Heidelberg (Other); Medical University of Vienna (Other); RWTH Aachen University (Other); Klinikum Arnsberg (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18524; 2019-001723-12 (EudraCT Number)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Venous Thromboses; Stent Stenosis
Keywords: Aspirin plus rivaroxaban vs. rivaroxaban for the prevention
MeSH Terms: conditions — Venous Thrombosis | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: a multi-center, international, randomized, open label, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin® (Experimental): To show if a combination therapy of rivaroxaban plus Aspirin® is more efficient (superiority testing) as rivaroxaban alone in the prevention of early venous stent thrombosis in patients suffering from post-thrombotic syndrome in the first 6 months following endovascular therapy.
  To demonstrate tolerability of combination therapy of Aspirin® plus rivaroxaban in long-term treatment.
  Interventions: Drug: Aspirin 100mg
- Control group (No Intervention): Observational study of standard of care anticoagulation (rivarobaban dosis defined in the clinical routine).

INTERVENTIONS:
Drug: Aspirin 100mg — Aspirin® cardio (CH) or Aspirin® protect (DE, AT) Film coated tablets Acetylsalicylic acid 100 mg Once daily oral intake for 6 months
  Other Names: Aspirin
  Arms: Aspirin®

SUMMARY:
To show if a combination therapy of rivaroxaban plus Aspirin® is more efficient (superiority testing) as rivaroxaban alone in the prevention of early venous stent thrombosis in patients suffering from post-thrombotic syndrome in the first 6 months following endovascular therapy To demonstrate tolerability of combination therapy of Aspirin® plus rivaroxaban in long-term treatment.

DETAILED DESCRIPTION:
Deep vein thrombosis is associated with severe morbidity and mortality. It is the most frequent type of venous thromboembolism (VTE) and responsible for approximately 800.000 deaths per year in the European Union and the United States combined. The post-thrombotic syndrome (PTS) is a frequent long-term complication of proximal deep vein thrombosis (DVT), which occurs in up to 50% of patients despite adequate anticoagulation therapy and compression stockings. Patients with DVT of the inferior vena cava or iliac veins are at highest risk for the development of PTS. Inadequate recanalization and persistent venous outflow obstruction promotes the development of venous hypertension, secondary valve damage, valvular reflux, and the clinical manifestation of PTS, which consists of a similar set of signs and symptoms as in superficial venous insufficiency. Symptoms may include leg edema, pruritus, dysesthesia, leg pain on standing, skin changes, venous claudication with limited exercise capacity, and leg ulcers. Venous ulcers occur in approximately 10% of patients with iliofemoral DVT after 3 years.

The diagnosis of PTS is made based on the presence of its clinical features, a prior history of proximal DVT, and the results of imaging studies. Clinical scores, such as the Villalta score, can function as a tool to stage severity of disease. PTS in classified as mild if the Villalta score is 5-9, moderate if the Villalta score is 10-14, and severe if the Villata score exceeds 15 points. Disabling venous claudication can be diagnosed by treadmill exercise tests. Magnetic resonance imaging venography can be used in addition to duplex ultrasound to objectify central venous obstruction, and unmark underlying strategic compression sides (e.g. May-Thurner syndrome).

Recommendations by the American Heart Association for endovascular treatment of PTS suggest percutaneous recanalization including the implantation of stents for symptomatic patients) Endovascular therapy with provisional stent placement shows promising clinical outcomes to improve PTS-associated symptoms, including leg ulcers. However, there is significant risk for early stent thrombosis, estimated as high as 21% after 12 months.

Antithrombotic therapy is the corner stone of the prevention of stent thrombosis, but there is great inconsistency in the use of antithrombotic agents. The value of extended anticoagulation therapy in PTS patients beyond the durations recommended in VTE management guidelines is controversial, and it has not been specifically investigated in the presence of venous stent implants. Although oral anticoagulants are accepted as the main therapy regimen, the benefit of antiplatelet therapy (APT) in the early phase after venous stent implantation is unclear.

According to a recent international survey completed by 106 experts, one third reported to use life-long anticoagulation with a vitamin-K antagonist (VKA), and another 19% chose life-long anticoagulation with direct anticoagulant (DOAC) for a presented case scenario of a PTS patients treated with venous stents. The use of APT following stent placement alone or in combination with an anticoagulant was reported in 7% and 13%, respectively, whereas 25% reported use of APT following discontinuation of ACT.

Conventionally, antiplatelet agents, such as acetylsalicylic acid, are regarded as drugs that prevent arterial thrombosis, as platelet adhesion predominates clotting in high-flow, high-sheer circulation.

There is compelling evidence that Aspirin® is effective in the prevention of arterial stent thrombosis, but it is unclear, whether it can prevent venous stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and data protection declaration obtained prior to any trial-specific procedures
2. Patient aged ≥18 years
3. Confirmed diagnosis of post-thrombotic syndrome defined as Villalta score > 4 points prior to enrolment and venous stent intervention
4. Confirmed stenosis of inferior vena cava, iliac vein, or common femoral vein by duplex ultrasound or cross-sectional imaging (CT venography or MR venography) prior to enrolment and venous stent intervention
5. Successfully conducted venous stent intervention involving either:

   * inferior vena cava
   * iliac vein or
   * common femoral vein
6. Patients either on active treatment with rivaroxaban or patients planned for treatment with rivaroxaban after intervention

Exclusion Criteria:

1. Previous venous intervention in target vessels
2. Any contraindication for antithrombotic therapy (e.g. active gastric ulcer, duodenal ulcer, bleeding disorder with increased tendency of bleedings)
3. Patients with a recent (3 months) clinically significant bleeding and / or active or recent (3 months) ulcerative or inflammatory gastrointestinal disease
4. Ongoing antiplatelet therapy or previous antiplatelet therapy within 7 days prior to Visit 1
5. Acute thrombosis (venous thromboembolism events < 3 months prior to Visit 1)
6. Pre-existing coagulopathy
7. Prior stroke or transient ischemic attack (< 12 months prior to Visit 1)
8. Pregnancy, breast feeding, or planned pregnancy within the trial period or women of childbearing potential not using an adequate method of contraception
9. Severe heart, liver or kidney disease
10. Severe somatopathic, neurological and / or psychiatric disease(s)
11. Malignant growth (concurrent or previous cancer with a relapse-free and treatment-free interval of less than 5 years before Visit 1)
12. Known hypersensitivity to acetylsalicylic acid (Aspirin® cardio or Aspirin® protect and / or its excipients), to other antiphlogistic drugs or to analgesics or anti-fever drugs
13. Concomitant intake of Methotrexat > 15 mg per week
14. Parallel participation in another clinical trial, participation in a clinical trial within less than 6 weeks prior to the Screening visit or previous participation in this clinical trial
15. Known to be, or suspected of being unable to comply with the trial protocol (e.g. no permanent address, history of drug abuse, known to be non-compliant or presenting an unstable psychiatric history)
16. Legal incapacity and / or other circumstances rendering the patient unable to understand the nature, scope and possible impact of the study
17. Custody by juridical or official order
18. Evidence of an uncooperative attitude
19. Difficulties in understanding the language in which the patient information is given
20. Patients dependent from the investigator or sponsor (e.g. close relatives of the investigator, employees of the clinic, the sponsor or involved CRO(s))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
The primary patency rate is defined as the percentage of patients with primary treatment success after 6 months | 6 month
  The primary patency rate is defined as the percentage of patients with primary treatment success after 6 months (=Visit 3), i.e. without the occurrence of either i) occlusion of at least a part of the stent segment or ii.) a re-intervention to maintain patency of the treated segment.

SECONDARY OUTCOMES:
Primary patency rate after 3 months | 3 month
  The primary patency rate is defined as the percentage of patients with primary treatment success after 3 months (=Visit 2), i.e. without the occurrence of either i) occlusion of at least a part of the stent segment or ii.) a re-intervention to maintain patency of the treated segment.
Secondary patency rate after 3 and 6 months | 3 and 6 months
  Secondary patency rate is defined as the percentage of patients with primary treatment success and without the occurrence of occlusion of at least a part of the stent segment, irrespective of any re-intervention
Primary sustained clinical success after 3 and 6 months (=Visit 2 and Visit 3) | 3 and 6 months
  Primary sustained clinical success, defined as the absence of post-thrombotic syndrome (Villalta score 0-4 points) without the need for repeated intervention assessed at the latest routine follow-up visit (at the latest available follow-up).
Difference between treatment groups in the incidence of patients with open stents but >50% residual stenosis according Duplex criteria | 3 month
  Difference between treatment groups in the incidence of patients with open stents but >50% residual stenosis according Duplex criteria
Difference of limb circumference | 3 and 6 months
  Difference of limb circumference of the affected leg in comparison to the contralateral leg at 3 and 6 months (= Visit 2 & 3), respectively, compared to baseline (for patients with only one affected leg)
Quality of life using the CIVIQ-20 (chronic venous insufficiency quality of life questionnaire) | 3 and 6 months
  Quality of life using the CIVIQ-20 (chronic venous insufficiency quality of life questionnaire) at 3 and 6 months (= Visit 2 & 3), respectively, compared to baseline.
  Value range: 20-100 points; Higher scores mean worse outcome
Change in Villalta score | 3 and 6 months
  Change in Villalta score with and without "ulcus cruris assessment" for the affected leg from baseline to 3 and 6 months (= Visit 2 & 3), respectively.
  Value range: 0-48 points; Higher scores mean worse outcome
Revised venous clinical severity score (rVCSS) | 3 and 6 months
  Revised venous clinical severity score (rVCSS) for the affected leg from baseline to 3 and 6 months (= Visit 2 & 3), respectively.
  Value range: 0-30 points; Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof.Dr.med., Study Chair — University Hospital, Zürich
Locations (6):
- Medizinische Universität Wien, Vienna, Austria
- Germany (4):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Klinikum Arnsberg - Karolinen Hospital, Arnsberg
  - Universitätsklinikum Freiburg, Bad Krozingen
  - Universitätsklinikum Heidelberg, Heidelberg
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barco S, Jalaie H, Sebastian T, Wolf S, Fumagalli RM, Lichtenberg M, Zeller T, Erbel C, Schlager O, Kucher N. Aspirin Plus Rivaroxaban Versus Rivaroxaban Alone for the Prevention of Venous Stent Thrombosis Among Patients With Post-Thrombotic Syndrome: The Multicenter, Multinational, Randomized, Open-Label ARIVA Trial. Circulation. 2025 Mar 25;151(12):835-846. doi: 10.1161/CIRCULATIONAHA.124.073050. Epub 2025 Jan 28. PMID 39874026